CLINICAL TRIAL: NCT03600649
Title: Phase 1 Trial of the LSD1 Inhibitor Seclidemstat (SP 2577) With and Without Topotecan and Cyclophosphamide in Patients With Relapsed or Refractory Ewing Sarcoma and Select Sarcomas
Brief Title: Clinical Trial of SP-2577 (Seclidemstat) in Patients With Relapsed or Refractory Ewing or Ewing-related Sarcomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Salarius Pharmaceuticals, LLC (Industry)
Collaborators: National Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SALA-002-EW16
Record Dates: First submitted 2018-06-04; First posted 2018-07-26 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Ewing Sarcoma; Myxoid Liposarcoma; Sarcoma,Soft Tissue; Desmoplastic Small Round Cell Tumor; Extraskeletal Myxoid Chondrosarcoma; Angiomatoid Fibrous Histiocytoma; Clear Cell Sarcoma; Primary Pulmonary Myxoid Sarcoma; Myoepithelial Tumor; Sclerosing Epithelioid Fibrosarcoma; Fibromyxoid Tumor
MeSH Terms: conditions — Sarcoma, Ewing; Liposarcoma, Myxoid; Sarcoma; Desmoplastic Small Round Cell Tumor; Chondrosarcoma, Extraskeletal Myxoid; Histiocytoma, Angiomatoid Fibrous; Sarcoma, Clear Cell; Myoepithelioma; Fibroma | interventions — seclidemstat; Cyclophosphamide; Topotecan

STUDY DESIGN:
Intervention Model Description: Two cohorts with single-agent seclidemstat in patients with myxoid liposarcoma and in patients with other sarcomas with similar chromosomal translocations to Ewing sarcoma (FET-family translocations), and one cohort of Ewing sarcoma patients treated with seclidemstat in combination with topotecan and cyclophosphamide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Myxoid Liposarcoma (Experimental): Twice-daily administration of oral seclidemstat
  Interventions: Drug: Seclidemstat
- Sarcomas with FET-family translocations, including demoplastic small round cell tumors (Experimental): Twice-daily administration of oral seclidemstat
  Interventions: Drug: Seclidemstat
- Ewing sarcoma, combination therapy (Experimental): Twice daily administration of seclidemstat in combination with cyclophosphamide and topotecan
  Interventions: Drug: Seclidemstat; Drug: Cyclophosphamide; Drug: Topotecan

INTERVENTIONS:
Drug: Seclidemstat — Twice daily administration of seclidemstat
  Other Names: LSD1 Inhibitor; SP-2577
Drug: Cyclophosphamide — 250 mg/m2/day on Days 1 thru 5 of a 21-day cycle
  Arms: Ewing sarcoma, combination therapy
Drug: Topotecan — 0.75 mg/m2/day on Days 1 thru 5 of a 21-day cycle
  Arms: Ewing sarcoma, combination therapy

SUMMARY:
Single agent, non-randomized, open label expansion in select sarcoma patients including myxoid liposarcoma and other sarcomas that share similar chromosomal translocations to Ewing sarcoma; AND dose expansion of the combination of seclidemstat with topotecan and cyclophosphamide in patients with Ewing sarcoma

DETAILED DESCRIPTION:
The single agent expansion cohort of select sarcoma patients will enroll myxoid liposarcoma patients and patients with other sarcomas that share similar chromosomal translocations to Ewing sarcoma (FET-family translocations), including but not limited to desmoplastic small round cell tumor.

A safety lead-in dose escalation and dose expansion will be conducted assessing the combination of seclidemstat with topotecan and cyclophosphamide in patients with relapsed or refractory Ewing sarcoma.

ELIGIBILITY:
Inclusion Criteria for All Patients

* Age ≥ 12 years and weight ≥ 40 kg.
* Karnofsky ≥ 70% for over ≥ 16 years old and Lansky ≥ 70% for under 16 years old, equivalent to Eastern Cooperative Oncology Group (ECOG) performance status Grade 0 or 1.
* Life expectancy of greater than 4 months in investigator's opinion.
* Willingness to provide tumor biopsies during screening and while on treatment. Optional for patients < 18 years of age and patients enrolled in the Ewing sarcoma combination treatment arm. Biopsies can be exempt if deemed by the investigator that the biopsy is not medically feasible for the patient or the patient is unfit for the procedure.
* Normal organ and marrow function as defined below:

  * absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * platelets ≥ 100 x 109/L; no transfusion 7 days prior to labs
  * total bilirubin ≤ 1.5 x upper limit of normal (ULN) or, in patients with Gilbert syndrome, total bilirubin > 1.5 x ULN as long as direct bilirubin is normal
  * AST and ALT ≤ 3 x ULN
  * creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above normal
* Ability to understand and the willingness to sign a written informed consent document.

Additional Inclusion Criteria for Ewing Sarcoma Combination Treatment Cohort

* Patients must have a histologic confirmed diagnosis of Ewing sarcoma with a known EWSR1 translocation through local assessment that is relapsed or refractory and must have received at least one prior course of therapy for Ewing sarcoma. For the purposes of this study, refractory disease is defined as metastatic or unresectable disease that has either progressed or is stable at completion of planned therapy.
* Patients must have had no more than 2 lines/courses of systemic treatment for Ewing sarcoma
* No prior therapy with the combination regimen of topotecan and cyclophosphamide. Prior cyclophosphamide is allowed if not combined with topotecan.
* Patients must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

Additional Inclusion Criteria for Single Agent Myxoid Liposarcoma Cohort and for Single Agent FET-Translocated Sarcomas

* Patients must have a histologic confirmed diagnosis of one of the following sarcomas that share similar known chromosomal translocations to Ewing sarcoma (per local assessment) and are relapsed or refractory and not amenable to surgery at time of enrollment.
* Patients must have received at least one prior course of systemic therapy but no more than 3 courses of systemic therapy for sarcoma.
* Patients must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

Exclusion Criteria for All Patients

* Patients who have not recovered to Grade 1 or baseline from adverse events related to prior therapy excluding lymphopenia, alopecia, peripheral neuropathy and ototoxicity, which are only exclusionary if original AE was ≥ CTCAE Grade 3.
* Patients receiving therapy with other anti-neoplastic or experimental agents.
* Prior therapy with LSD1 targeted agents including monoamine oxidases for cancer therapy.
* Prior oral tyrosine kinase inhibitors (i.e. sorafenib, pazopanib, regorafenib, cabozantanib) within 14 days of Cycle 1 Day 1.
* Other, prior systemic anti-cancer treatment (chemotherapy or biologic therapy [i.e. monoclonal antibodies]) within 21 days prior to Cycle 1 Day 1. For agents that have known adverse events occurring beyond 21 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Medical Monitor.
* Prior therapy with immunotherapy such as a checkpoint inhibitor, cellular therapy or vaccine therapy within 28 days prior to Cycle 1 Day 1. Patients must have recovered from any immune-related adverse events to Grade 1 or baseline and require ≤ 10 mg of prednisone equivalent daily. Patients with immune-related hypothyroidism and/or hypoadrenalism may enroll while on thyroid or hydrocortisone replacement therapy, respectively.
* Prior small port palliative radiotherapy within 14 days of Cycle 1 Day 1 or within 42 days of Cycle 1 Day 1 from definitive local control radiation (any dose greater than 50 Gy, within 42 days of Cycle 1 Day 1).
* Prior therapy with long acting myeloid growth factor within 14 days of Cycle 1 Day 1 or within 7 days of Cycle 1 Day 1 from a short acting myeloid growth factor.
* Evidence of graft versus host disease or prior allo- or auto-bone marrow transplant or stem cell infusion within 84 days from Cycle 1 Day 1 or receiving immunosuppressants following a stem cell procedure.
* Participation in a prior investigational study within 30 days prior to Cycle 1 Day 1 or within 5 half-lives of the investigational product, whichever is longer.
* Progressive or symptomatic brain metastases; patients with brain metastases may be included in this trial as long as the brain metastases have received definitive treatment and are stable (i.e., no evidence of progression). The brain metastases must be stable for a minimum of 6 weeks prior to Cycle 1 Day 1.
* Currently receiving any of the following substances and cannot be discontinued 14 days or 5 half-lives for CYP inhibitors (whichever is shorter) prior to Cycle 1 Day 1:

  * moderate or strong inhibitors or inducers of major CYP isoenzymes, including grapefruit, grapefruit hybrids, pomelos, star fruit, and Seville oranges
  * moderate or strong inhibitors or inducers of major drug transporters
  * substrates of CYP3A4/5 with a narrow therapeutic index
* Uncontrolled concurrent illness including, but not limited to:

  * ongoing or active infection
  * transfusion dependent thrombocytopenia or anemia
  * psychiatric illness/social situations that would limit compliance with study requirements; discuss with Medical Monitor if there are any questions
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

  * symptomatic congestive heart failure
  * left ventricular ejection fraction (LVEF) ≤ 50%
  * unstable angina pectoris or cardiac arrhythmia
  * baseline QTc (Fridericia) ≥ 450 milliseconds
  * long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome
* Any major surgery within 21 days prior to Cycle 1 Day 1. Major surgery is defined as any significantly invasive procedure into a major body cavity (abdomen, cranium etc.) and/or surgery requiring extensive recuperation (joint replacement). Please discuss with Medical Monitor if there are any questions.
* Pregnant and breastfeeding women are excluded from this study. The effects of seclidemstat on the developing human fetus have the potential for teratogenic or abortifacient effects.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of seclidemstat administration.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with seclidemstat. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of seclidemstat (SP-2577) as a single agent and in combination with topotecan and cyclophosphamide measured by dose limiting toxicities and adverse events according to CTCAE version 5.0 | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To evaluate the safety and tolerability of seclidemstat (SP-2577) as a single agent and in combination with topotecan and cyclophosphamide in patients with relapsed or refractory Ewing sarcoma and select sarcomas. Toxicities will be graded in severity per the guidelines outlined in the NCI CTCAE version 5.0. The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which ≥ 2 patients from a cohort of 3 to 6 patients experience a dose-limiting toxicity.

SECONDARY OUTCOMES:
Determine the maximum tolerated dose of SP-2577 as determined by dose limiting toxicities measured according to CTCAE version 5.0 | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To determine the maximum tolerated dose (MTD) of seclidemstat as a single agent and in combination with topotecan and cyclophosphamide in patients with relapsed or refractory Ewing sarcoma. Toxicities will be graded in severity per the guidelines outlined in the NCI CTCAE version 5.0. The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which ≥ 2 patients from a cohort of 3 to 6 patients experience a dose-limiting toxicity.
Characterization of the pharmacokinetics of SP-2577 as measured by peak plasma concentration | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To characterize pharmacokinetics of seclidemstat as a single agent and in combination with topotecan and cyclophosphamide.
Characterization of the pharmacokinetics of SP-2577 as measured by area under the curve | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To characterize pharmacokinetics of seclidemstat as a single agent and in combination with topotecan and cyclophosphamide.
Characterization of the pharmacokinetics of SP-2577 as measured by apparent clearance of seclidemstat | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To characterize pharmacokinetics of seclidemstat as a single agent and in combination with topotecan and cyclophosphamide.
Characterization of the pharmacokinetics of SP-2577 as measured by median half-life | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To characterize pharmacokinetics of seclidemstat as a single agent and in combination with topotecan and cyclophosphamide.
Food effects on the pharmacokinetics of SP-2577 as measured in both fasted and fed populations, primarily measured by apparent clearance. | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To evaluate the effect of food on the pharmacokinetics of seclidemstat. Both fasted and fed PK samples will be taken.
Anti-tumor activity as measured according to RECIST 1.1 criteria based upon radiological assessments. | From screening through at least 30 days after end of treatment, up to approximately 24 months
  To evaluate the anti-tumor activity of seclidemstat as a single agent and in combination with topotecan and cyclophosphamide. Tumor response will be measured according to RECIST 1.1 criteria. Radiological assessments may be centrally collected and subjected to quality checks and review by a central imaging vendor at the discretion of Salarius.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Mayo Clinic, Jacksonville, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington, Seattle, Washington